CLINICAL TRIAL: NCT02035735
Title: Usefulness of Narrow-band Imaging to Estimate the Superficial Spread of Squamous Cell Carcinomas in Oropharynx, Hypopharynx and Larynx
Brief Title: Interest of Narrow Band Imaging in Detection of Upper Aerodigestive Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13 203 02
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Squamous Cell Carcinoma of Oropharynx; Squamous Cell Carcinoma of Hypopharynx; Squamous Cell Carcinoma of Larynx
Keywords: NBI,; squamous cell carcinoma,; pharynx, larynx, surgical margins.
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell; Laryngeal Diseases; Margins of Excision | interventions — Narrow Band Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Videoendoscopy with WL and NBI (Experimental): The day before the laryngoscopy under general anesthesia (LGA), two endoscopies by two different physicians were performed for each patients and recorded: the first one with white light (WL) and the second one with NBI (NBI).
  Interventions: Procedure: WL and NBI

INTERVENTIONS:
Procedure: WL and NBI — For each patient with a suspicion of squamous cell carcinoma of the oropharynx, hypopharynx or larynx for whom a laryngoscopy under general anesthesia (LGA) is expected benefit the day before a transnasal endoscopy with white lamp (WL) and NBI by two different operators. Suspected mucosal abnormalities showed by one or the two technics are reported in a table wich describes the different areas of the pharynx and the larynx. During the LGA, several biopsies are performed and identified (WL and/or NBI).

SUMMARY:
The aim of this study is to prospectively determine if the use of NBI endoscopy modifies the superficial extension of these tumors.

DETAILED DESCRIPTION:
Several studies have already showed the interest of the use of NBI for the early diagnosis of malignancies of the upper aerodigestive tract. For all tumors, the most accurate evaluation of its limits is very important to perform the best strategy of treatment. If surgery seems to be the best option, surgical margins must be widely healthy. Despite the systematic transnasal flexible endoscopy with white lamp followed by laryngoscopy under general anesthesia (LGA) and tomodensitometric evaluation, surgical margins can be unhealthy (in situ carcinoma or dysplasia). We propose to evaluate if the use of the NBI could be useful to determine the superficial spread of squamous cell carcinomas in these locations.

To April 2013 to Mars 2015, all patients with a suspicion of squamous cell carcinoma of the oropharynx, hypopharynx or larynx and whom a LGA are expected, are included. The day before the LGA, two endoscopies by two different physicians were performed for each patients and recorded: the first one with white light and the second one with NBI. All results are noted on a schema. Superficial extension or synchronous lesions showed by NBI are analysed and compared with with lamp technic.

After surgery, surgical margins were evaluated and healthy margins were measured.

ELIGIBILITY:
Inclusion Criteria:

- Patients who can benefit a laryngoscopic exam under general anesthesia

Exclusion Criteria:

* General anesthesia contra-indications
* Local anesthesia allergy
* Breast-feeding period or pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of patients for whom superficial extension of the tumors has been increased by NBI. | 4 minutes

SECONDARY OUTCOMES:
Number of tumors upstaged. | 4 minutes
Contribution of the NBI in the diagnosis of other synchronous locations. | 4 minutes
Contribution of the NBI in the diagnosis of pre-neoplastic lesions. | 4 minutes
Contribution of the NBI in the evaluation of surgical margins. | 4 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien VERGEZ, MD, PhD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chabrillac E, Espinasse G, Lepage B, Uro-Coste E, Dupret-Bories A, De Bonnecaze G, Vergez S. Contribution of narrow band imaging in delineation of laryngopharyngeal superficial cancer spread: a prospective study. Eur Arch Otorhinolaryngol. 2021 May;278(5):1491-1497. doi: 10.1007/s00405-020-06499-2. Epub 2021 Jan 5. PMID 33398548